CLINICAL TRIAL: NCT05605821
Title: Influence of Diabetic Control on the Degree of Liver Fibrosis Assessed by Non-invasive Scores in Patients Followed in Diabetology: a Retrospective Study
Brief Title: Influence of Diabetic Control on the Degree of Liver Fibrosis Assessed by Non-invasive Scores in Patients Followed in Diabetology
Acronym: DIAFIB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DIAFIB
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic steatopathy (nonalcoholic fatty liver disease or NAFLD) has seen its prevalence soar in recent years that it is now the leading cause of chronic liver disease in developed countries, surpassing viral and alcoholic etiologies and affecting approximately 25% of the world's population. This growth is explained by a change in eating habits, lifestyle, and the increase in the prevalence of obesity in the general population. This hepatopathy evolves in successive stages in a slow and insidious manner: from simple fatty overload in the liver (NALF, steatosis), to steatosis plus hepatic inflammation (NASH - "nonalcoholic steatohepatitis"), up to the stage of cirrhosis with all its own complications Isolated steatosis has a rather benign course, whereas the transition to NASH is associated with a high risk of general mortality and liver-related causes. NASH is the stage at which fibrogenesis accelerates with the risk of progression to cirrhosis and/or primary liver cancer. The degree of hepatic fibrosis has a major influence on the prognosis of patients with NAFLD. Specifically, the presence of fibrosis greater than or equal to 2 (F≥2) is associated with increased risk of liver events and liver-related mortality. The risk of cardiovascular events increases as early as fibrosis grade 1 (F≥1). In addition, the presence of advanced fibrosis or cirrhosis (F≥3) greatly increases the risk of developing hepatocellular carcinoma, and patients require biannual monitoring by liver ultrasound. Systematic screening of diabetic patients with advanced fibrosis is necessary to establish specific surveillance. Non-invasive scores have been developed to assess the degree of liver fibrosis in patients with NAFLD. Among these scores, FIB4 ("Score Fibrosis-4") has the advantage of being easy to use in routine practice with good diagnostic performance for liver fibrosis in patients with NAFLD. A FIB4 value ≤ 1.3 has a negative predictive value of 90% for the diagnosis of severe fibrosis (F≥3), whereas a FIB4 > 2.67 has a positive predictive value of 80% for severe fibrosis. Diagnostic performance is poorer for patients older than 65 years, and an FIB4 cutoff <2 is used in this case to identify those at very low risk of advanced fibrosis. This score is calculated from platelet count, patient age, and transaminases (ASAT: Aspartate-Amino-Transferase and ALAT: Alanine-Amino-Transferase) according to the following formula: (age x ASAT) / (platelets x √[ALAT]). It allows selection of patients with a higher risk of advanced fibrosis who will require further investigations and specialist advice. It also allows to avoid unnecessary explorations in patients with a low risk of advanced fibrosis (FIB4<1.3 if age<65 years or FIB4<2 if age>65 years). There is currently no pharmacological treatment with market authorization. The mainstay of treatment is a change in lifestyle and habits (dietary and behavioral, including increased physical activity) with the aim of "fat cleansing" the liver. There is a strong link between the presence of type 2 diabetes and the risk of developing NAFLD and/or NASH. NAFLD is present in 70% of patients with type 2 diabetes. Furthermore, the presence of diabetes is associated with an increased risk of developing advanced fibrosis, cirrhosis and hepatocellular carcinoma in patients with NAFLD. Glycation end products are substances that result from the reaction between a carbohydrate and protein residues, but can also result from lipid oxidation. These molecules have been associated with accelerated aging and increased risk of cardiovascular disease. The accumulation of glycation end products during periods of prolonged hyperglycemia seems to contribute to the progression of hepatic fibrosis. In this context, our study aims to evaluate the impact of type 2 diabetes control on the degree of liver fibrosis using non-invasive tests. The primary objective is to evaluate the association between diabetic disease control and the degree of liver fibrosis. The secondary objectives are: to evaluate the practices in terms of evaluation of hepatic fibrosis and management of diabetic patients at risk of advanced fibrosis in a tertiary diabetes service, to evaluate the association between the use of certain treatments and the degree of hepatic fibrosis, to evaluate the impact of the variation of the Body Mass Index (BMI) on hepatic fibrosis and to evaluate the percentage of patients at risk of severe fibrosis in a population of type 2 diabetic patients followed up in a tertiary diabetology service.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥ 18 years
* Patient with a diagnosis of type 2 diabetes, identified by ICD-10 codes, among patients hospitalized between 01/03/2018 and 17/03/2020 in HDJ in the Diabetes Service of GHPSJ
* French-speaking patient

Exclusion Criteria:

* Absence of at least one HbA1c measurement per year available over a period of 5 years (This is obtained by different means: handwritten in the patient's file, performed in the HDJ, performed in town and integrated into the patient's file, reported orally by the patient during the follow-up consultation. Glycated hemoglobin data for the 5-year retrospective period available).
* Lack of sufficient data to calculate the non-invasive fibrosis score FIB4.
* Secondary diabetes (neoplasia, chronic calcifying pancreatitis, post pancreatectomy pancreatic insufficiency for various reasons: see figure 8 below)
* HDJ for pre-bariatric surgery evaluation
* Other declared causes of chronic liver disease according to the patient's medical record
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosis of type 2 diabetes, identified by ICD-10 codes, among patients hospitalized between 01/03/2018 and 17/03/2020 in HDJ in the Diabetes Service of GHPSJ.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the association between diabetic disease control and the degree of hepatic fibrosis | Month1
  This outcome corresponds to the level of association between long-term diabetes control estimated from the evolution of glycated hemoglobins (HbA1c) over the study period and the degree of liver fibrosis assessed by the FIB4 score (non-severe fibrosis: FIB4<1.3 if age<65 years or FIB4<2 if age>65 years; severe or undetermined fibrosis: FIB4>1.3 if age<65 years or FIB4>2 if age>65 years).

SECONDARY OUTCOMES:
Practices in terms of evaluation of hepatic fibrosis and management of patients | Month 1
  This outcome corresponds to the percentage of patients at risk of advanced fibrosis who had additional investigations (pulse elastometry, liver biopsy) and were referred to hepatology.
Association between the use of certain treatments and the degree of hepatic fibrosis | Month1
  This outcome corresponds to the association between the use of antidiabetic treatments and the degree of hepatic fibrosis.
Impact of Body Mass Index (BMI) variation on liver fibrosis | Month1
  This outcome corresponds to the BMI value at study entry and the degree of fibrosis according to the FIB4 score at entry and its evolution over time.
Percentage of patients at risk of severe fibrosis in a population of type 2 diabetics followed in a tertiary diabetes service. | Month1
  This outcome corresponds to the percentage of patients with severe fibrosis in a population of type 2 diabetics.

CONTACTS AND LOCATIONS:
Overall Officials: Adela VOICAN, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Hôpital Antoine Béclert, Clamart
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Younossi ZM, Stepanova M, Afendy M, Fang Y, Younossi Y, Mir H, Srishord M. Changes in the prevalence of the most common causes of chronic liver diseases in the United States from 1988 to 2008. Clin Gastroenterol Hepatol. 2011 Jun;9(6):524-530.e1; quiz e60. doi: 10.1016/j.cgh.2011.03.020. Epub 2011 Mar 25. PMID 21440669
- [Background] Torres DM, Williams CD, Harrison SA. Features, diagnosis, and treatment of nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2012 Aug;10(8):837-58. doi: 10.1016/j.cgh.2012.03.011. Epub 2012 Mar 23. PMID 22446927
- [Background] McPherson S, Hardy T, Dufour JF, Petta S, Romero-Gomez M, Allison M, Oliveira CP, Francque S, Van Gaal L, Schattenberg JM, Tiniakos D, Burt A, Bugianesi E, Ratziu V, Day CP, Anstee QM. Age as a Confounding Factor for the Accurate Non-Invasive Diagnosis of Advanced NAFLD Fibrosis. Am J Gastroenterol. 2017 May;112(5):740-751. doi: 10.1038/ajg.2016.453. Epub 2016 Oct 11. PMID 27725647
- [Background] Hamaguchi E, Takamura T, Sakurai M, Mizukoshi E, Zen Y, Takeshita Y, Kurita S, Arai K, Yamashita T, Sasaki M, Nakanuma Y, Kaneko S. Histological course of nonalcoholic fatty liver disease in Japanese patients: tight glycemic control, rather than weight reduction, ameliorates liver fibrosis. Diabetes Care. 2010 Feb;33(2):284-6. doi: 10.2337/dc09-0148. Epub 2009 Oct 30. PMID 19880582
- See also: Related Info — https://www.fmcgastro.org/texte-postu/postu-2019-paris/nash-recommandations-easl-2017/